CLINICAL TRIAL: NCT07308236
Title: An Open-Label, Single Dose Study to Determine the Metabolism and Excretion of [14C]E2086 in Healthy Male Participants
Brief Title: A Study to Determine the Metabolism and Excretion of [14C]E2086 in Healthy Male Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: E2086-A001-004
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- E2086 (Experimental)
  Interventions: Drug: E2086

INTERVENTIONS:
Drug: E2086 — E2086 oral capsule.

SUMMARY:
The primary purpose of this study is to determine the metabolism and excretion of [14C]E2086 in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking and non-vaping, healthy male, age greater than or equal to (>=) 18 years and less than or equal to (<=) 55 years old at the time of informed consent
2. Body Mass Index (BMI) >=18 and less than (<) 30 kilogram per square meter (kg/m^2) at Screening
3. Provide written informed consent
4. Willing and able to comply with all aspects of the protocol

Exclusion Criteria:

1. Have previously been dosed in more than 2 radiolabeled drug studies in the past 12 months. For participants who have previously been dosed in 2 or more radiolabeled drug studies within the last 12 months, the previous radiolabeled dose must be at least 4 months prior to check-in to the trial site where exposures are known to the investigator, or 6 months prior to check-in to the trial site for a radiolabeled drug trial where exposures are not known to the investigator. The total 12-month exposure from this trial and a maximum of 2 other previous radiolabeled studies must be within the CFR recommended levels considered safe, per US Title 21 CFR 361.1.
2. Exposure to significant diagnostic or therapeutic radiation (eg, serial x-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to check-in.
3. Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners must meet the following criteria: not of childbearing potential or practicing highly effective contraception throughout the trial period and for 28 days after trial drug discontinuation. No sperm donation is allowed during the trial period and for 90 days after trial drug discontinuation.

   NOTE: All female partners of male participants will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing). Examples of highly effective contraception include total abstinence, an intrauterine device, a double-barrier method (such as condom plus diaphragm with spermicide), a contraceptive implant, and oral contraceptive. Female partners of male participants who have not had a successful vasectomy, who use hormonal contraception, must be on the same hormonal contraceptive for 28 days before the male participants are dosed with trial drug, throughout the trial period and for 28 days afterwards.
4. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing.
5. Evidence of disease that may influence the outcome of the trial within 4 weeks before dosing, eg, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, orbcardiovascular system.
6. Any history of surgery that may affect PK profiles of E2086 (eg, hepatectomy, nephrectomy, digestive organ resection) or participants who have a congenital abnormality in metabolism at Screening.
7. Any clinically abnormal symptom or organ impairment found by medical history at Screening, and physical examinations, vital signs, electrocardiogram (ECG) findings, or laboratory test results that require medical treatment at Screening or Baseline.
8. Initiation of statin therapy, or a change to a different statin, or an increase in the dose of a statin within the 6 months before the planned start of the study
9. A prolonged QT/QTc interval (QTcF greater than (>) 450 millisecond [ms]) as demonstrated by the mean of triplicate ECGs (recorded at least 1 min apart) at Screening or Baseline
10. Systolic blood pressure >130 millimeter of mercury (mmHg) or diastolic blood pressure >85 mmHg at Screening or Baseline
11. Heart rate <50 beats/min or >100 beats/min at Screening or Baseline
12. Any lifetime history of suicidal ideation or any lifetime history of suicidal behavior as indicated by the Columbia-Suicide Severity Rating Scale (C-SSRS).
13. Any lifetime history of psychiatric disease (including, but not limited to, depression or other mood disorders, bipolar disorder, psychotic disorders, including schizophrenia, panic attacks, and anxiety disorders [if ever treated with medication]).
14. Known history of clinically significant drug allergy at Screening or Baseline
15. Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening or Baseline.
16. Known to be human immunodeficiency virus (HIV) positive at Screening
17. History of drug or alcohol dependency or abuse within the 2 years before Screening, or those who have a positive urine drug test or alcohol test at Screening or Baseline.
18. Currently enrolled in another clinical trial or used any investigational drug or device within 30 days (or 5 half-lives, whichever is longer) preceding informed consent
19. Use of illegal recreational drugs and marijuana
20. Receipt of blood products within 4 weeks, or donation of blood within 8 weeks, or donation of plasma within 1 week before dosing.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-02-23 (Estimated)

PRIMARY OUTCOMES:
Mass Balance Recovery of E2086, Expressed as Cumulative Percent of the Radiolabeled Dose | Day 1 up to Day 21
  Mass balance will be determined by pharmacokinetic (PK) analysis of [14C]E2086 and E2086 in the biological matrices.
Maximum Observed Concentration (Cmax) of [14C]E2086 for Total Radioactivity (TRA) in Plasma | Day 1 up to Day 21
Time to Reach Cmax (Tmax) of [14C]E2086 for TRA in Plasma | Day 1 up to Day 21
Area Under the Concentration-time Curve from Zero Time to Time of Last Quantifiable Concentration [AUC (0-t)] of [14C]E2086 for TRA in Plasma | Day 1 up to Day 21
Area Under the Concentration-time Curve from Zero Time Extrapolated to Infinite Time [AUC (0-inf)] of [14C]E2086 for TRA in Plasma | Day 1 up to Day 21
Terminal Elimination Phase Half-life (t1/2) of [14C]E2086 for TRA in Plasma | Day 1 up to Day 21
Cmax of [14C]E2086 for TRA in Whole Blood | Day 1 up to Day 21
Tmax of [14C]E2086 for TRA in Whole Blood | Day 1 up to Day 21
AUC (0-t) of [14C]E2086 for TRA in Whole Blood | Day 1 up to Day 21
AUC (0-inf) of [14C]E2086 for TRA in Whole Blood | Day 1 up to Day 21
t1/2 of [14C]E2086 for TRA in Whole Blood | Day 1 up to Day 21
Cmax of E2086 and its Metabolite M1 in Plasma Using liquid Chromatography Coupled With Mass Spectrometry (LC-MS/MS) | Day 1 up to Day 21
Tmax E2086 and its Metabolite M1 in Plasma Using LC-MS/MS | Day 1 up to Day 21
AUC (0-t) of E2086 and its Metabolite M1 in Plasma Using LC-MS/MS | Day 1 up to Day 21
AUC (0-inf) of E2086 and its Metabolite M1 in Plasma Using LC-MS/MS | Day 1 up to Day 21
t1/2 of E2086 and its Metabolite M1 in Plasma Using LC-MS/MS | Day 1 up to Day 21
Apparent Total Clearance (CL/F) of E2086 in Plasma Using LC-MS/MS | Day 1 up to Day 21
Apparent Volume of Distribution (Vz/F) at Terminal Phase of E2086 in Plasma Using LC-MS/MS | Day 1 up to Day 21
Metabolite Ratio (MRp) of E2086 and its Metabolite M1 in Plasma Using LC-MS/MS | Day 1 up to Day 21
Cumulative Amount Excreted in Urine from Zero Time to Time of Last Interval (Ae) of E2086 and its Metabolite M1 in Urine Using LC-MS/MS | Day 1 up to Day 21
Fraction of Dose Excreted in Urine from Zero Time to Time of Last Interval (Fe) of E2086 and its Metabolite M1 in Urine Using LC-MS/MS | Day 1 up to Day 21
Renal Clearance (CLR) of E2086 and its Metabolite M1 in Urine Using LC-MS/MS | Day 1 up to Day 21
MRu of E2086 and its Metabolite M1 in Urine Using LC-MS/MS | Day 1 up to Day 21
Percentage of Administered Radioactive Dose Excreted in Urine, Feces, and Toilet Tissue by TRA | Day 1 up to Day 21

SECONDARY OUTCOMES:
Characterization of Metabolites in Plasma, Urine, Feces After Administration of a Single Oral Dose of Radiolabeled [14C]E2086 | Up to 70 days
  Metabolite profiling in plasma, urine, and feces will be performed by radio-high performance liquid chromatography (HPLC) methods and/or accelerator mass spectrometry. Metabolites (M1) and other metabolites will be identified and estimated on the radiochromatograms, and the amount of each metabolite will be quantified based on the peak areas on the radiochromatograms. For metabolites detected on the radiochromatograms, LC-MS/MS analysis may be performed to estimate and identify their chemical structures.
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to 70 days
Number of Participants With Abnormal Laboratory Parameter Values | Up to 70 days
Number of Participants With Clinically Significant Change in Vital Sign Values | Up to 70 days
Number of Participants With Clinically Significant Change in 12-Lead Electrocardiogram (ECG) Values | Up to 70 days

CONTACTS AND LOCATIONS:
Locations (1):
- Fortrea Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.